CLINICAL TRIAL: NCT03088189
Title: Effect of Parental Peri-conceptional Vitamin B12 Supplementation on Infant Neurocognitive Development in Offspring
Status: Terminated | Type: Observational
Why Stopped: Assessments were stopped in February 2020 due to COVID pandemic
Sponsor: Kem Hospital, Pune, India (Other)
Responsible Party: Principal Investigator, Dr. Chittaranjan S Yajnik, Director, Diabetes Unit, Kem Hospital, Pune, India
Other Study IDs: KEMHRC/ADHOC/25
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Neurodevelopmental Disorders
Keywords: maternal nutrition; periconceptional; neurocognitive development
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vitamin B12 group: Mothers in the group are receiving vitamin B12 2µg supplements daily
- Multiple micronutrient group: mothers in this group are receiving vitamin B12 2µg plus multiple micronutrients (MMN) plus 20g of milk powder
- Placebo: Mothers are receiving placebo

SUMMARY:
Maternal nutrition is an important factor which determines fetal growth and development. Micronutrients vitamin B12 and folic acid are essential determinants of one carbon metabolism and play an important role in DNA synthesis, methylation and epigenetic regulation of gene expression. Diabetes unit of KEMHRC, Pune has been conducting the Pune Rural Intervention in Young Adolescents since last 3 years. Subjects of the PMNS cohort have been randomized as part of a controlled trial of nutritional intervention with vitamin B12 vs multiple micronutrient and milk protein vs placebo. This study aims to understand the intergenerational effects of vitamin B12 supplementation. 74 infants have been born in this trial since 2013. This study would assess neurocognitive development of offspring born to mothers who are part of the nutritional intervention trial; on the Bayley scales of infant and toddler development - III. The study aims to test the hypothesis that infants born to mothers who received vitamin B12 would have favorable infant neurocognitive development scores as compared to placebo. And this effect would be enhanced in the group whose mothers received MMN with milk protein.

DETAILED DESCRIPTION:
Background:

The concept of fetal programming suggests that adverse intrauterine growth environment influences development of fetal organ structure and function, hence laying the basis for risk for chronic disease in later life with its consequent effects on human capital. One of the important factors determining intrauterine growth is maternal and fetal nutritional status. Micronutrients vitamin B12 and folic acid are essential determinants of one carbon metabolism and play an important role in DNA synthesis, methylation and epigenetic regulation of gene expression. The ongoing Pune Maternal Nutritional Study (PMNS) has demonstrated an association between low maternal vitamin B12 levels during pregnancy and impaired cognitive functioning in offspring at 9 and 12 years of age. This observation suggests that maternal micronutrient status during pregnancy can influence neurocognitive development and functioning in later life. Various other intervention studies conducted in Delhi and Bangladesh support that vitamin B12 and folic acid supplementation in children between 6-30 months of age can improve their motor and neurocognitive development. On this background the Diabetes unit of KEMHRC, Pune has been conducting the Pune Rural Intervention in Young Adolescents since last 3 years. Subjects of the PMNS cohort have been randomized as part of a controlled trial of nutritional intervention with vitamin B12 vs multiple micronutrient and milk protein vs placebo. This study aims to understand the intergenerational effects of vitamin B12 supplementation. 74 infants have been born in this trial since 2013. This presents a unique opportunity to study the effects of parental periconceptional vitamin B12 supplementation on infant neurocognitive development.

Objective and Hypothesis:

To compare group differences, in infant neurocognitive development scores assessed at 24 months of age between mothers who received either vitamin B12 alone, or MMN with milk protein or placebo.

Hypothesis: Infants born to mothers who received vitamin B12 would have favorable infant neurocognitive development scores as compared to placebo. And this effect would be enhanced in the group whose mothers received MMN with milk protein.

Methods:

Study subjects:

The study subjects will include infants born to parents who are enrolled in the PRIYA trial. As of August 2016, 74 infants have been born in the trial the oldest being born in June 2013. The subject recruitment will be ongoing and any infants born subsequently will also be included.

Procedure:

After institutional and ethical clearance, parents of infants approaching 24 months of age would be approached for study and informed consent obtained from the parents. The infant with parent would be brought to KEM hospital after scheduling an appointment. Assessment Bayley scales of infant and toddler development - III would be performed at the TDH center of KEM hospital by a trained assessor. All assessments would be performed at age of 24±2 months. For infants who are already older than 24 months assessment would be performed at their current age after obtaining approval for the study from the institutional ethics committee.

Tool:

The Bayley scales of infant and toddler development - III is a standardized instrument for assessing motor and neurocognitive development in infants. The scale assess development on the domains of cognitive, receptive communication, expressive communication, fine motor, gross motor, socio-emotional. The scale provides a general adaptive composite score along with scores on the individual domains.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born to parent enrolled in the PRIYA trial
2. Age > 24 months and < 48 months
3. Informed consent obtained from parents

Exclusion Criteria:

1. Infants diagnosed to have known genetic syndromes with mental retardation or cerebral palsy
2. Infants with recent immunization or febrile illness will be assessed 1 week after resolution

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children born to mothers who are part of an ongoing nutritional intervention trial. Mothers are randomised to receive either Vitamin B12, B12 with multiple micronutrients and milk protein or placebo
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Composite cognitive score and subdomain scores on Bayley scales of infant and toddler development - III | assessed at 2 years of age
  Scores obtained on the assessment scale would be compared between groups

SECONDARY OUTCOMES:
Total score on Child Behavior Check list | assessed at 2 years of age
  Scores obtained on the assessment scale would be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Chittaranjan Yajnik, MD, Principal Investigator — KEM Hospital research center, Pune
Locations (1):
- Diabetes Unit, Kem Hospital Research Centre, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official webpage of diabetes unit KEM hospital research center Pune — http://kemdiabetes.org